CLINICAL TRIAL: NCT01590901
Title: The Pharmacokinetics and Safety Study of Probucol by Multiple Administration in Healthy Male Subjects
Brief Title: Pharmacokinetics and Safety Study of Probucol by Multiple Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 009-11-803-01
Record Dates: First submitted 2012-01-11; First posted 2012-05-03 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Probucol; healthy male subjects
MeSH Terms: interventions — Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- probucol in healthy male subjects (Other): multiple oral doses of probucol in single group of healthy male subjects
  Interventions: Drug: Probucol

INTERVENTIONS:
Drug: Probucol — 250mg (1 tablet) bid. p.o for 14 consecutive days
  Other Names: Lorelco

SUMMARY:
The Objectives of this study is to evaluate the pharmacokinetics and safety of multiple oral doses of probucol in healthy male subjects.

DETAILED DESCRIPTION:
This is a single dose, single period, multiple administration, open-labeled trial in one investigation center.

The screening examination will be completed from Day -14 to Day -2 before investigational medicinal product (IMP) administration. The subjects will be hospitalized on Day -1. From Day 1 (the next day), the subjects will receive probucol twice daily (BID). for 14 consecutive days. On Day 18, the subjects can be discharged after the safety evaluation. The follow-up visit will occur on Day 6, 9, 12, 15, 19, 27 (totally 41 days) after the final dosing day.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese.
2. Gender: Male.
3. Age 20 to 40 years, (at time of informed consent).
4. Body mass index [BMI, body weight (kg) / height (m)2] between 19 and 26 kg/m2, inclusive.
5. Nonsmokers (or former smokers): Urinary cotinine level satisfying the criteria for a nonsmoker established by the trial site (at time of screening examination).
6. Subjects judged by the investigator to be healthy based on the medical history, physical examination, vital signs, 12 lead ECG, the results of serological test (HIV/HCV Ab, HBsAg and Syphilis Ab) and clinical laboratory tests, etc.

Exclusion Criteria:

1. Subjects with hypersensitivity or a history of hypersensitivity to any drug (any prescription or over-the-counter [OTC] drug)
2. Subjects who meet any of the following lipid criteria in the fasting state (at time of screening examination)

   * LDL-C: ≥ 140 mg/dL
   * TC: ≥ 220 mg/dL
   * HDL-C: < 40 mg/dL
   * TG: ≥ 150 mg/dL

     * LDL-C value will be directly measured or calculated by the Friedewald formula. Friedewald Formula: LDL-C = TC - HDL-C - TG/5 (When TG value is less than 400 mg/dL) LDL-C value will be directly measured when TG value is 400 mg/dL or greater.
3. Subjects with electrocardiogram (ECG) results showing AV block or with both QTc and QRS width outside the standard values of the ECG laboratory (at time of screening examination)
4. Subjects with alcohol or drug dependence or a history of drug abuse
5. Subjects who have a positive result in an infectious disease test or urine drug test (at time of screening examination)
6. Use of any of the following within the specified period prior to scheduled investigational medicinal product (IMP) administration

   * All other prescription and OTC drugs (within 2 weeks prior to scheduled IMP administration)
   * Alcohol and caffeine-containing products (within 1 week prior to scheduled IMP administration)
7. Use of any other investigational drug within 16 weeks prior to scheduled IMP administration in the present trial
8. Plasmapheresis or plateletpheresis within 2 weeks or whole blood collection (blood donation, etc) cumulatively exceeding 200 mL within 4 weeks, 400 mL within 12 weeks, or 1200 mL within 1 year prior to scheduled IMP administration
9. Subjects whose body weight is less than 50 kg (at time of screening examination)
10. Subjects who are scheduled for examination or treatment at any other hospital or clinic during the trial period
11. Subjects otherwise judged by the investigator or sub investigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Day 1, 3, 5, 7, 9, 11, 12, 13, 14
  Pharmacokinetic parameters:
  Day 1 (Plasma PK parameters over the 24h dosing period)： Cmax, Cmax1, Cmax2, tmax1, tmax2, AUC (0-10)h, AUC (10-24)h, AUC24h, C24h; Day3，5，7，9，11，12，13：C24h; Day 14： Cmax, Cmax1, Cmax2, tmax1, tmax2, AUC (0-10)h, AUC (10-24)h, AUC24h, C24h, Clast, tlast, t1/2,z,Lambdaz, DF, CL/F, Vz/F, AUC_%Extrap;
  Accumulation evaluation parameters:
  Rpred, R14,ac(AUC24h), R14,ac(Cmax), R14,ac(C24h), R14,ac[AUC(0-10h)], R14,ac[AUC(10-24h)], R14,ac(Cmax1), R14,ac(Cmax2).

CONTACTS AND LOCATIONS:
Overall Officials: Pei Hu, PHD, Principal Investigator — Clinical Pharmacology Research Center of Peking Union Medical College Hospital
Locations (1):
- Clinical Pharmacology Research Center, Peking Union Medical College Hospital, Beijing, China